CLINICAL TRIAL: NCT05452928
Title: Aciclovir for HSV-2 Meningitis: A Double-blind Randomised Controlled Trial (AMEN)
Brief Title: Aciclovir Versus Placebo for HSV-2 Meningitis
Acronym: AMEN
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jacob Bodilsen (Other)
Responsible Party: Sponsor-Investigator, Jacob Bodilsen, Sponsor-investigator, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMEN1; 2020-000033-41 (EudraCT Number)
Record Dates: First submitted 2022-07-01; First posted 2022-07-12 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Herpes Simplex 2; Meningitis, Viral
Keywords: meningitis; HSV-2; Herpes simplex 2; viral meningitis; aseptic meningitis; acyclovir; valacyclovir; aciclovir; valaciclovir
MeSH Terms: conditions — Meningitis, Viral; Meningitis; Meningitis, Aseptic | interventions — Acyclovir; Valacyclovir

STUDY DESIGN:
Intervention Model Description: Investigator initiated, double-blind, 2-arm (1:1 allocation), international, multicentre, parallel group, randomised, placebo controlled, superiority trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: We will use a centralised internet-based computer-generated randomisation schedule prepared and overseen by an experienced statistician. Patients will be randomised in a 1:1 ratio in permuted blocks of two to six and stratified by country, sex, and adjunctive dexamethasone treatment (yes/no).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active arm (Active Comparator): Randomisation to 7 days of active treatment with IV aciclovir 10 mg/kg q8h and possibility for oral step-down therapy with valaciclovir 1g q8h, or placebo (IV q8h and/or oral q8h).
  Interventions: Drug: Acyclovir 50 MG/ML
- Placebo (Placebo Comparator): Randomisation to 7 days of IV and/or oral placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acyclovir 50 MG/ML — Patients are randomised to active treatment with IV acyclovir with the possibility of step-down to valacyclovir. If the treating physician prefers, initial IV treatment can be omitted and the patient can be treated with valacyclovir throughout the study period.
  Other Names: Valacyclovir
  Arms: Active arm
Drug: Placebo — Placebo either in IV formulation or as tablets identical to valacyclovir tablets.
  Arms: Placebo

SUMMARY:
To determine whether active treatment with (val)acyclovir is superior for treatment of viral meningitis compared with placebo assessed by numbers meeting a primary, objective endpoint at 7 days after randomisation

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age admitted on suspicion of viral meningitis defined as:

  1. A clinical presentation consistent with viral meningitis (e.g. headache, nuchal rigidity, photophobia, or fever) AND
  2. Cerebrospinal fluid (CSF) pleocytosis (>4 leukocytes x 106/L) AND
  3. HSV-2 positive by PCR of the CSF
  4. Glasgow Coma Scale score of 15 AND
  5. Ability to absorb oral medications

Exclusion Criteria:

* Patients fulfilling any of the following criteria will be excluded:

  1. Encephalitis as defined by the International Encephalitis Consortium if diagnosed during standard care (see Glossary)20
  2. Transverse myelitis as defined by the Transverse Myelitis Consortium Working Group if diagnosed during standard care (see Glossary)21
  3. Severe immuno-compromise defined as an ongoing need for biological- or chemotherapy (e.g. natalizumab), prednisolone >20 mg/day for ≥14 days, uncontrolled HIV/AIDS (see glossary), haematological malignancies, and organ transplant recipients14,18,22
  4. Moderate to severe concomitant genital herpes requiring systemic aciclovir
  5. Pregnancy (proven by positive urine or plasma human chorionic gonadotropin test in fertile women)
  6. Hepatic impairment (aspartate aminotransferase or alanine aminotransferase levels >5 times the upper limit of normal)
  7. Impaired renal function (estimated glomerular filtration rate <25 mL/min)
  8. Intolerance to (val)aciclovir
  9. Probenecid treatment
  10. Systemic antiviral therapy with an antiherpetic effect for >24 hours
  11. Previous enrolment into this trial

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint (proportion with a Total Morbidity Score) | 7 days since randomisation
  The proportion with a Total Morbidity Score (TMS) >6 is considered treatment failure. The score is a sum of scores for headache (range 0 to 6), nuchal rigidity (range 0 to 4), photophobia (range 0 to 4), myalgia (range 0 to 4), fever (range 0 to 4), nausea (range 0 to 4). The score thus ranges from 0 to 21 with higher scores indicating more severe symptoms.

SECONDARY OUTCOMES:
Secondary endpoint 1 (Proportion of patients with ≤50% reduction of Total Morbidity Score) | 7 days since randomisation
  Proportion of patients with ≤50% reduction of Total Morbidity Score since randomisation. Please see characterization of score under primary endpoint.
Secondary endpoint 2 Extended Glasgow outcome scale score | 7 days, 3 months, and 12 months since randomisation
  Extended Glasgow outcome scale score. Range 1 to 8 with higher scores indicating better outcome.
Secondary endpoint 3 All-cause mortality | 7 days, 3 months, and 12 months since randomisation
  All-cause mortality
Secondary endpoint 4 EQ-5D-5L | 7 days, 3 months, and 12 months since randomisation
  EQ-5D-5L. Comprises 5 questions with an ordinal scale from 1 to 5 with higher scores indicating more morbidity. Finally, a visual analog score is filled ranging from 0 to 100 with higher scores indicating better health.
Secondary endpoint 5 Mental Fatigue Scale | 7 days, 3 months, and 12 months since randomisation
  Mental Fatigue Scale. Comprises 14 questions with scores from 0 to 3 with higher values suggesting more morbidity. A combined score >10.5 usually suggests mental fatigue problems.
Secondary endpoint 6 (SF-36) | 7 days, 3 months, and 12 months since randomisation
  Short Form Health Survey 36 (SF-36). Scores eight different domains from 0 to 100 with higher values indicating no disability.
Secondary outcome 7 neurological deficit | 7 days, 3 months, and 12 months since randomisation
  Any new neurological deficit reported by patient or observed during clinical examination
Secondary outcome 8 Completion of assigned treatment | 7 days since randomisation
  Completion of assigned treatment (active or placebo) assessed by administered intravenous or oral treatment as signed off by nurses in hospitalized patients and pill counts for patients discharged with oral study drug.
Secondary outcome 9 complications | 7 days since randomisation
  Peripheral venous line associated complications (i.e. catheter-associated infection, thrombosis, or haemorrhage).
Secondary outcome 10Severe adverse events | 7 days since randomisation
  Severe adverse events, i.e. incident treatment-emergent serious adverse events.

IPD SHARING:
Plan to Share IPD: Yes
Data will be deposited at Mendeley Data (https://data.mendeley.com/).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning six months and ending three years after publication, an anonymized dataset can be shared.
Access Criteria: Qualified researchers who provide a methodologically sound proposal.
URL: https://data.mendeley.com/